CLINICAL TRIAL: NCT06819436
Title: Effect of Dexamethasone on Post-spinal Hypotension in Geriatric Patients Undergoing Orthopaedic Surgery at Tertiary Care Hospital Karachi.
Brief Title: Effect of Dexamethasone on Post-spinal Hypotension
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shaheed Mohtarma Benazir Bhutto Institue of Trauma (Other)
Responsible Party: Principal Investigator, Maria Shafi, Principal Investigator, Shaheed Mohtarma Benazir Bhutto Institue of Trauma
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ERC-000105/SMBBIT/2023; Not funded (Other Grant/Funding Number: SMBBIT)
Record Dates: First submitted 2025-02-05; First posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Post Spinal Anaesthesia Hypotension; Geriatric Population; Orthopedic Surgeries
MeSH Terms: interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexamethasone Group (Experimental): Participants randomly allocated to this group will receive intravenous dexamethasone 8mg preoperatively 20 minutes before spinal anesthesia
  Interventions: Drug: Dexamethasone
- Placebo Group (Placebo Comparator): Participants randomly allocated to this group will receive placebo preoperatively 20 minutes before spinal anesthesia
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Dexamethasone — Intravenous dexamethasone 8mg given to participants before spinal anesthesia
  Arms: Dexamethasone Group
Other: Placebo — Intravenous placebo given to the participants before spinal anesthesia
  Arms: Placebo Group

SUMMARY:
The goal of this clinical trial is to learn if intravenous dexamethasone is effective for prevention of post spinal hypotension in geriatric population undergoing orthopedic surgeries. The main question aim to answer is:

Does intravenous dexamethasone in participants undergoing orthopedic procedures of lower limb under spinal anesthesia prevents post spinal hypotension? Researchers are comparing two groups of participants

* Participants in (Dexamethasone Group) Group D are receiving intravenous dexamethasone 8mg preoperatively
* Participants in (Placebo Group) Group P are receiving placebo preoperatively.

ELIGIBILITY:
Inclusion Criteria:

Patient undergoing orthopedic surgery in spinal anesthesia. ASA ≤ 2.

Exclusion Criteria:

Patients with history of cardiac arrhythmias. Patients with history of acute coronary syndrome. Patient with history of polytrauma. Patients with contraindication to SA (e.g., coagulopathy, thrombocytopenia, allergy to local anesthetic agent) and those on steroids or serotonin related medications (e.g., selective serotonin reuptake inhibitor) will be excluded.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Post spinal Anesthesia Hypotension | From enrollment to 30 minutes after spinal anesthesia
  Hypotension will be considered if there will be 25% decrease below the baseline for (Mean Arterial Pressure) MAP and will be managed by 300 ml of (Normal Saline) NS solution with incremental intravenous 5 mg doses of ephedrine. The proportion of patients with hypotension at any time during the first 20 min after induction of the (Spinal Anesthesia) SA and before starting the surgical procedure will be considered as the outcome of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Shaheed Mohtarma Benazir Bhutto Institute of Trauma, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided